CLINICAL TRIAL: NCT05724485
Title: Effect of Branched-chain Amino Acids (BCAA) to Muscle Cramps in Patients With Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Watcharasak Chotiyaputta, Associate professor, Faculty of Medicine, Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 1071/2020
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Muscle Cramp; Cirrhosis; Quality of Life
Keywords: Muscle Cramp; cirrhosis
MeSH Terms: conditions — Muscle Cramp; Fibrosis | interventions — Amino Acids, Branched-Chain; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will be randomized to receive BCAA or placebo. The BCAA and placebo were prepared by pharmacists who contained both 12.45 grams of BCAA and placebo in the same quantity, the same containing sachet, and labeled enveloped from No.1 to No.50. The sequence of labels was randomized by computer generator block of 4 randomizations with conceal allocation to investigators, participants, care providers, and outcomes assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCAA group (Active Comparator): 12.45 grams of branched-chain amino acids orally per day before bedtime for 12 weeks.
  Interventions: Drug: Branched-chain Amino Acid
- Placebo group (Placebo Comparator): 12.45 grams of placebo (Maltodextrin) orally per day before bedtime for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Branched-chain Amino Acid — 12.45 grams of BCAA orally per day before bedtime
  Arms: BCAA group
Drug: Placebo — 12.45 grams of Maltodextrin orally per day before bedtime
  Other Names: Maltodextrin
  Arms: Placebo group

SUMMARY:
The goal of this randomized controlled trial is to compare the efficacy and safety of branched-chain amino acids (BCAA) versus placebo for treating muscle cramps in cirrhotic patients. The main questions it aims to answer are:

* Compared the effect of BCAA versus placebo on muscle cramp frequency in cirrhotic patients
* Compared the effect of BCAA versus placebo on muscle cramp duration and severity in cirrhotic patients
* Compared the effect of BCAA versus placebo on quality of life in cirrhotic patients with muscle cramps Participants with cirrhosis who have experienced muscle cramps at least once per week will be randomized to receive either a placebo or 12.45 grams of BCAA orally per day for 12 weeks.

DETAILED DESCRIPTION:
Cirrhosis is a late-stage of fibrosis of the liver caused by many forms of liver disease. Muscle cramps are visible or palpable involuntary contraction part of the muscle. The prevalence of cramps in cirrhosis varied range from 31-78%. The pathophysiology of cramps in cirrhosis was explained by multiple mechanisms such as energy metabolism, nerve function, and plasma volume. Cramps significantly diminished the quality of life in cirrhotic patients.

Many drugs, vitamins, and minerals were studied for treating cramps in cirrhosis in previous studies but no clinical improvement, good randomized control studies, or side effects.

Branched-chain amino acids (BCAA) had been developed to correct this amino acid imbalance and helped to decrease the frequency of cramps and improve the quality of life in cirrhotic patients from previous studies but there were no control groups and a small number of patients were included. The aim of this study was to evaluate the efficacy and safety of BCAA for controlling muscle cramps in cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Muscle cramp ≥ 1 time per week
* Confirmed cirrhotic status (radiologic finding compatible with cirrhosis or liver stiffness measurement ≥ 12.5 kPa by transient elastography method or pathological confirm of cirrhosis)

Exclusion Criteria:

* Allergy to BCAA
* Overt hepatic encephalopathy
* Hepatorenal syndrome
* Severe renal insufficiency; eGFR < 30
* Heart failure
* Peripheral arterial disease
* Active malignancies beyond hepatocellular carcinoma
* Heavy alcohol drinking (> 21g/day for men and >14g/day for women)
* Pregnancy or lactation
* Current use of BCAA within 3 months
* Recent adding or titrating diuretics within 4 weeks
* On current medications for muscle cramp relief such as vitamin E, taurine, carnitine, narcotic pain medications, baclofen, methocarbamol, other muscle relaxers, NSAIDs, or other antispastic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change of muscle cramp frequency | 12 weeks
  Change from baseline in muscle cramp frequency by patient's diary record

SECONDARY OUTCOMES:
Change of muscle cramp duration | 12 weeks
  Change from baseline in muscle cramp duration by patient's diary record as minutes per muscle cramp events
Change of muscle cramp severity | 12 weeks
  Change from baseline in muscle cramp severity by patient's diary record as the visual analog scale that reported from 0 (no pain) to 10 (worst pain).
Quality of life in cirrhotic patients with muscle cramps | 12 weeks
  Change of quality of life in cirrhotic patients with muscle cramps at the end of the study compared to baseline by chronic liver disease questionnaire (CLDQ) that includes 29 items in the following domains: abdominal symptoms, fatigue, systemic symptoms, activity, emotional function, and worry. The response of CLDQ results in 1 to 7 scales: ranging from "all of the time" to "none of the time".
Muscle mass in cirrhotic patients with muscle cramps | 12 weeks
  Change of muscle mass in cirrhotic patients with muscle cramps at the end of the study compared to baseline by bioelectrical impedance analysis (BIA)
Muscle strengthening in cirrhotic patients with muscle cramps | 12 weeks
  Change of muscle strength in cirrhotic patients with muscle cramps at the end of the study compared to baseline by hand grip strength measurement
Serum albumin | 12 weeks
  Change of serum albumin (g/dL) in cirrhotic patients with muscle cramps at the end of the study compared to baseline
Serum alanine aminotransferase | 12 weeks
  Change of serum alanine aminotransferase in cirrhotic patients with muscle cramps at the end of the study compared to baseline
Serum aspartate aminotransferase | 12 weeks
  Change of serum aspartate aminotransferase in cirrhotic patients with muscle cramps at the end of the study compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Siwaporn Chainuvati, Asso Prof, Principal Investigator — 66643249159
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chatrath H, Liangpunsakul S, Ghabril M, Otte J, Chalasani N, Vuppalanchi R. Prevalence and morbidity associated with muscle cramps in patients with cirrhosis. Am J Med. 2012 Oct;125(10):1019-25. doi: 10.1016/j.amjmed.2012.03.012. Epub 2012 Jul 24. PMID 22835465
- [Result] Mehta SS, Fallon MB. Muscle cramps in liver disease. Clin Gastroenterol Hepatol. 2013 Nov;11(11):1385-91; quiz e80. doi: 10.1016/j.cgh.2013.03.017. Epub 2013 Mar 28. PMID 23542334
- [Result] Soeters PB, Fischer JE. Insulin, glucagon, aminoacid imbalance, and hepatic encephalopathy. Lancet. 1976 Oct 23;2(7991):880-2. doi: 10.1016/s0140-6736(76)90541-9. PMID 62115
- [Result] Vidot H, Carey S, Allman-Farinelli M, Shackel N. Systematic review: the treatment of muscle cramps in patients with cirrhosis. Aliment Pharmacol Ther. 2014 Aug;40(3):221-32. doi: 10.1111/apt.12827. Epub 2014 Jun 18. PMID 24942957
- [Result] Sako K, Imamura Y, Nishimata H, Tahara K, Kubozono O, Tsubouchi H. Branched-chain amino acids supplements in the late evening decrease the frequency of muscle cramps with advanced hepatic cirrhosis. Hepatol Res. 2003 Aug;26(4):327-329. doi: 10.1016/s1386-6346(03)00152-9. PMID 12963433
- [Result] Hidaka H, Nakazawa T, Kutsukake S, Yamazaki Y, Aoki I, Nakano S, Asaba N, Minamino T, Takada J, Tanaka Y, Okuwaki Y, Watanabe M, Shibuya A, Koizumi W. The efficacy of nocturnal administration of branched-chain amino acid granules to improve quality of life in patients with cirrhosis. J Gastroenterol. 2013 Feb;48(2):269-76. doi: 10.1007/s00535-012-0632-x. Epub 2012 Jul 24. PMID 22825550
- [Result] Sobhonslidsuk A, Silpakit C, Kongsakon R, Satitpornkul P, Sripetch C. Chronic liver disease questionnaire: translation and validation in Thais. World J Gastroenterol. 2004 Jul 1;10(13):1954-7. doi: 10.3748/wjg.v10.i13.1954. PMID 15222044
- [Result] Arguedas MR, DeLawrence TG, McGuire BM. Influence of hepatic encephalopathy on health-related quality of life in patients with cirrhosis. Dig Dis Sci. 2003 Aug;48(8):1622-6. doi: 10.1023/a:1024784327783. PMID 12924658
- [Result] Younossi ZM, Guyatt G, Kiwi M, Boparai N, King D. Development of a disease specific questionnaire to measure health related quality of life in patients with chronic liver disease. Gut. 1999 Aug;45(2):295-300. doi: 10.1136/gut.45.2.295. PMID 10403745
- [Result] Kawaguchi T, Izumi N, Charlton MR, Sata M. Branched-chain amino acids as pharmacological nutrients in chronic liver disease. Hepatology. 2011 Sep 2;54(3):1063-70. doi: 10.1002/hep.24412. Epub 2011 Jun 23. PMID 21563202
- [Result] Abd-Elsalam S, Arafa M, Elkadeem M, Elfert A, Soliman S, Elkhalawany W, Badawi R. Randomized-controlled trial of methocarbamol as a novel treatment for muscle cramps in cirrhotic patients. Eur J Gastroenterol Hepatol. 2019 Apr;31(4):499-502. doi: 10.1097/MEG.0000000000001310. PMID 30444744
- [Result] Elfert AA, Abo Ali L, Soliman S, Zakaria S, Shehab El-Din I, Elkhalawany W, Abd-Elsalam S. Randomized placebo-controlled study of baclofen in the treatment of muscle cramps in patients with liver cirrhosis. Eur J Gastroenterol Hepatol. 2016 Nov;28(11):1280-4. doi: 10.1097/MEG.0000000000000714. PMID 27467714
- [Result] Nakaya Y, Okita K, Suzuki K, Moriwaki H, Kato A, Miwa Y, Shiraishi K, Okuda H, Onji M, Kanazawa H, Tsubouchi H, Kato S, Kaito M, Watanabe A, Habu D, Ito S, Ishikawa T, Kawamura N, Arakawa Y; Hepatic Nutritional Therapy (HNT) Study Group. BCAA-enriched snack improves nutritional state of cirrhosis. Nutrition. 2007 Feb;23(2):113-20. doi: 10.1016/j.nut.2006.10.008. PMID 17234504
- [Result] Marchesini G, Bianchi G, Merli M, Amodio P, Panella C, Loguercio C, Rossi Fanelli F, Abbiati R; Italian BCAA Study Group. Nutritional supplementation with branched-chain amino acids in advanced cirrhosis: a double-blind, randomized trial. Gastroenterology. 2003 Jun;124(7):1792-801. doi: 10.1016/s0016-5085(03)00323-8. PMID 12806613
- [Result] Muto Y, Sato S, Watanabe A, Moriwaki H, Suzuki K, Kato A, Kato M, Nakamura T, Higuchi K, Nishiguchi S, Kumada H; Long-Term Survival Study Group. Effects of oral branched-chain amino acid granules on event-free survival in patients with liver cirrhosis. Clin Gastroenterol Hepatol. 2005 Jul;3(7):705-13. doi: 10.1016/s1542-3565(05)00017-0. PMID 16206505
- [Result] Angeli P, Albino G, Carraro P, Dalla Pria M, Merkel C, Caregaro L, De Bei E, Bortoluzzi A, Plebani M, Gatta A. Cirrhosis and muscle cramps: evidence of a causal relationship. Hepatology. 1996 Feb;23(2):264-73. doi: 10.1002/hep.510230211. PMID 8591851
- [Result] Marchesini G, Bianchi G, Amodio P, Salerno F, Merli M, Panella C, Loguercio C, Apolone G, Niero M, Abbiati R; Italian Study Group for quality of life in cirrhosis. Factors associated with poor health-related quality of life of patients with cirrhosis. Gastroenterology. 2001 Jan;120(1):170-8. doi: 10.1053/gast.2001.21193. PMID 11208726
- [Result] Ng K, Lin CS, Murray NM, Burroughs AK, Bostock H. Conduction and excitability properties of peripheral nerves in end-stage liver disease. Muscle Nerve. 2007 Jun;35(6):730-8. doi: 10.1002/mus.20765. PMID 17387740
- [Result] Gluud LL, Dam G, Les I, Marchesini G, Borre M, Aagaard NK, Vilstrup H. Branched-chain amino acids for people with hepatic encephalopathy. Cochrane Database Syst Rev. 2017 May 18;5(5):CD001939. doi: 10.1002/14651858.CD001939.pub4. PMID 28518283
- [Result] Ko CH, Wu SJ, Wang ST, Chang YF, Chang CS, Kuan TS, Chuang HY, Chang CM, Chou W, Wu CH. Effects of enriched branched-chain amino acid supplementation on sarcopenia. Aging (Albany NY). 2020 Jul 26;12(14):15091-15103. doi: 10.18632/aging.103576. Epub 2020 Jul 26. PMID 32712600
- [Result] Sawada Y, Shiraki M, Iwasa M, Hiraoka A, Nakanishi H, Karino Y, Nakajima T, Miyaaki H, Kawaguchi T, Yoshiji H, Okita K, Koike K. The effects of diuretic use and the presence of ascites on muscle cramps in patients with cirrhosis: a nationwide study. J Gastroenterol. 2020 Sep;55(9):868-876. doi: 10.1007/s00535-020-01694-8. Epub 2020 Jun 12. PMID 32533302
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. J Hepatol. 2018 Aug;69(2):406-460. doi: 10.1016/j.jhep.2018.03.024. Epub 2018 Apr 10. No abstract available. PMID 29653741
- [Result] Angeli P, Fasolato S, Mazza E, Okolicsanyi L, Maresio G, Velo E, Galioto A, Salinas F, D'Aquino M, Sticca A, Gatta A. Combined versus sequential diuretic treatment of ascites in non-azotaemic patients with cirrhosis: results of an open randomised clinical trial. Gut. 2010 Jan;59(1):98-104. doi: 10.1136/gut.2008.176495. PMID 19570764